CLINICAL TRIAL: NCT02110836
Title: The Impact of Sucrose Ingestion During Exercise on Liver and Muscle Glycogen Concentration.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Gonzalez, PhD (Other)
Collaborators: University of Newcastle Upon-Tyne (Other); Maastricht University (Other); Sugar Nutrition, UK (Unknown)
Responsible Party: Sponsor-Investigator, Javier Gonzalez, PhD, Research Fellow, Northumbria University
Organization: Northumbria University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NUSUCA
Record Dates: First submitted 2014-04-03; First posted 2014-04-10 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Liver and Muscle Glycogen Use During Exercise.

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose ingestion (Active Comparator): Glucose ingestion during exercise at a rate of 1.8 g/min.
  Interventions: Dietary Supplement: Glucose ingestion
- Sucrose ingestion (Experimental): Sucrose ingestion during exercise at a rate of 1.8 g/min.
  Interventions: Dietary Supplement: Sucrose ingestion

INTERVENTIONS:
Dietary Supplement: Glucose ingestion — Glucose ingestion during exercise at 1.8 g/min
  Arms: Glucose ingestion
Dietary Supplement: Sucrose ingestion — Sucrose ingestion during exercise at 1.8 g/min
  Arms: Sucrose ingestion

SUMMARY:
Carbohydrate is stored in the body as glycogen, which is mainly found in the liver and muscle. During endurance exercise, muscle glycogen is used as fuel for the working muscles and liver glycogen is broken down to provide glucose to maintain blood glucose (sugar) levels. Both liver and muscle glycogen are important for the ability to perform intense/prolonged endurance exercise. Therefore, nutritional strategies which can maximise the availability of glycogen in muscle and liver can benefit endurance exercise capacity.

The carbohydrates typically found in sports drinks are glucose and sometimes fructose. If glucose only is ingested during exercise, then the maximum rate at which can be absorbed from the intestine into the blood stream is ~1 g/min. However, if different sources of carbohydrate (fructose) are used, which are absorbed through a different pathway, absorption of carbohydrate can be up to ~1.8 g/min. With more carbohydrate available as a fuel, this translates into an improvement in performance.

Sucrose is a naturally occurring sugar that is made up of a single glucose and single fructose molecule. Therefore, theoretically, this can use the two different pathways of absorption and also maximise carbohydrate delivery. It is not yet known however, what impact this has on our liver and muscle glycogen stores during exercise. Therefore the aim of this study is to assess whether sucrose ingestion influences liver and muscle glycogen depletion during endurance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18 - 35 years of age
* Endurance trained cyclist/triathlete
* VO2 max ≥ 50 ml/kg/min

Exclusion Criteria:

* Use of medication
* Smoking
* Metabolic disorders

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in liver glycogen concentration | 3 hours
  The change in liver glycogen concentration will be determined pre-to-post 3 h of exercise using 13C magnetic resonance spectroscopy.

SECONDARY OUTCOMES:
Plasma glucose concentration. | 3 hours
  Plasma glucose concentrations will be determined every 30 min during 3 h of exercise.
Plasma lactate concentration | 3 hours
  Plasma lactate concentrations will be determined every 30 min during 3 h of exercise.
Plasma non-esterified fatty acid concentration | 3 hours
  Plasma non-esterified fatty acid concentrations will be determined every 30 min during 3 h of exercise.
Indirect calorimetry | 3 hours
  Measurements of oxygen consumption, carbon dioxide production and respiratory exchange ratio through indirect calorimetry measured every 30 minutes during exercise.
Muscle glycogen concentration | 3 hours
  The change in muscle glycogen concentration will be determined pre-to-post 3 h of exercise using 13C magnetic resonance spectroscopy.
Change in intramyocellular lipid concentration | 3 hours
  The change in intramyocellular lipid concentration will be determined pre-to-post 3 h of exercise using 1H magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Gonzalez JT, Fuchs CJ, Smith FE, Thelwall PE, Taylor R, Stevenson EJ, Trenell MI, Cermak NM, van Loon LJ. Ingestion of glucose or sucrose prevents liver but not muscle glycogen depletion during prolonged endurance-type exercise in trained cyclists. Am J Physiol Endocrinol Metab. 2015 Dec 15;309(12):E1032-9. doi: 10.1152/ajpendo.00376.2015. Epub 2015 Oct 20. PMID 26487008